CLINICAL TRIAL: NCT02617303
Title: Effectiveness of an Intervention Through Physical Exercise for the Prevention of Falls and Its Consequences in Elderly People (75-89 Years) Performed in Primary Care: Study Protocol for a Randomized Controlled Trial
Brief Title: Prevention of Falls and Its Consequences in Elderly People
Acronym: PRECIOSA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P14/099
Record Dates: First submitted 2015-06-11; First posted 2015-11-30 (Estimated); Last update posted 2021-06-22 (Actual); Status verified 2020-10

CONDITIONS: Accidental Falls; Osteoporosis
Keywords: elderly; accidental falls; osteoporosis; fractures; Primary Care; Randomized clinical trial; Otago exercise programme
MeSH Terms: conditions — Osteoporosis; Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OTAGO'S program arm (Experimental): Patients meeting the inclusion criteria will be randomly assigned to the experimental group. They will receive OTAGO'S exercise program during three months, followed by adherence phase. Falls and fractures will be quarterly followed during 15 months.
  Interventions: Procedure: OTAGO's exercises
- CONTROL GROUP (Active Comparator): Patients meeting the inclusion criteria will be randomly assigned to the control group. Normal medical treatment will be provided by family physicians and nurses. Falls and fractures will be quarterly followed during 15 months.
  Interventions: Procedure: COMMON PRACTICE

INTERVENTIONS:
Procedure: OTAGO's exercises — The intervention is based on OTAGO's program, consisting of a set of aerobic exercises affecting gait, balance, stability and are adapted for older people to support them both in groups and individually. The program lasts 6 weeks (2 sessions per week) and is followed by a loyalty phase to consolidate the exercise program. Falls and fractures will be monitored quarterly for 15 months.
  Arms: OTAGO'S program arm
Procedure: COMMON PRACTICE — Normal medical treatment will be provided by family physicians and nurses.
  Arms: CONTROL GROUP

SUMMARY:
Falls are an important risk factor for fragility fractures. Both are associated with the ageing process and as they rise also increase the risk of mortality, disability and dependency. Interventions to prevent falls have been based on multifactorial approaches but the outcomes have shown little effectiveness. Lately, it is being recommended interventions which foster physical exercise incorporating it to daily life activities. The OTAGO exercise programme is based on easy physical exercises for older adults and has shown cost-effective outcomes for falls prevention and its consequences.

DETAILED DESCRIPTION:
This is a randomized clinical trial carried out in primary care. The study's scope of activity will include ten urban primary care centers. All selected patients with inclusion criteria will receive a geriatric assessment and other required medical treatment. Next, they will be allocated either to an intervention group or control group. The intervention group will be trained for three months according to the OTAGO exercise program (training phase). Followed by a loyalty phase during which they will be monitored quarterly for a year by their assessment team. The control group will be receive normal medical treatment. Falls and fractures will be monitored quarterly in both groups during 15 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 75 to 89 years at baseline assigned to Primary Care Team and living in the community
* Ranking the Folstein Mini Mental State Examination test
* Expectation of permanence in the area at least 18 months.
* Agree to participate in the study by informed consent, after reading the patient information sheet.

Exclusion Criteria:

* Current participation in another trial or institutional program of guided physical activity.
* Patients with who have had a hip and/or knee operation or major injury or any other intervention in the last 6 months.
* Patients with who are unable to follow an aerobic physical activity program. Patients using assisted mobility devices are not excluded.
* Patients in Home Care Programs or Nursing Homes at baseline or during the training phase.
* Terminal or severe cancer cases.
* Patients disabled prior to or during the study period.
* Have not been visited in reference's Health Center in the last two years (displacement / transfer
* Very advanced dementia that not allows to follow the instructions in the exercise program and nurse's instructions. In case of a caregiver who assume the realization of exercise program and the following of tips, it may be included.
* Displaced, will temporarily shifted (>2months/year) o will definitively shifted patients of Health Center.

Ages: 75 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 402 (Estimated)
Dates: Start 2015-09; Primary Completion 2019-09 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Reduction of falls measured with a questionnaire from April 2016 to June 2017. | 15 months
  Evaluate the incidence of OTAGO's physical intervention program on fall reduction in elderly (75-89years). Starting training with phase guided by physiotherapist, followed by loyalty phase guided by regular nurse. It will be measured with a questionnaire at baseline and during follow-up.

SECONDARY OUTCOMES:
Reduction of fracture measured with a questionnaire (location, causes and consequences) from April 2016 to June 2017. | 15 months
  Evaluate the incidence of OTAGO's physical intervention program on fracture reduction in elderly (75-89years). Starting training with phase guided by physiotherapist, followed by loyalty phase guided by regular nurse. It will be measured with a questionnaire (location, causes and consequences) at baseline and during follow-up.
Reduction of fear to fall measured with Falls Efficacy Scale (FES) from April 2016 to June 2017. | 15 months
  Evaluate the incidence of OTAGO's physical intervention program on reduction of fear to fall in elderly (75-89years). Starting training with phase guided by physiotherapist, followed by loyalty phase guided by regular nurse. It will be measured with Falls Efficacy Scale (FES) at baseline and during follow-up.
Parameters of physical frailty (strength) measured with switched test Timed Get Up and Go (TGUAG) from April 2016 to June 2017. | 15 months
  Evaluate the incidence of OTAGO's physical intervention program on improvement of parameters of physical frailty (strength) in elderly (75-89years). Starting training with phase guided by physiotherapist, followed by loyalty phase guided by regular nurse. It will be measured with switched test Timed Get Up and Go (TGUAG) at baseline and during follow-up.
Parameters of physical frailty (balance) measured through Biodex Balance System ('stability index') from April 2016 to June 2017. | 15 months
  Evaluate the incidence of OTAGO's physical intervention program on improvement of parameters of physical frailty (balance) in elderly (75-89years). Starting training with phase guided by physiotherapist, followed by loyalty phase guided by regular nurse. It will be measured through Tinneti Scale and Biodex Balance System. Biodex Balance System provides valid, reliable and repeatable objective measures of a patient's ability to balance on stable and unstable surfaces. It provides visual biofeedback of a patient's ability to control their centre of gravity and their limits of stability. This test provides an objective 'stability index' that if higher than the predicted value indicates a strength, proprioception, and vestibular or visual impairment. Both monitoring at baseline and during follow-up.
Parameters of physical frailty (motion) measured through "BTS G-WALK" from April 2016 to June 2017. | 15 months
  Evaluate the incidence of OTAGO's physical intervention program on improvement of parameters of physical frailty (flexibility) in elderly (75-89years). Starting training with phase guided by physiotherapist, followed by loyalty phase guided by regular nurse. It will be measured through "BTS G-WALK". It is a wireless laptop, its software allows to analyze basic parameters of motion. It will be monitoring at baseline and during follow-up.
Parameters of physical frailty (endurance) measured with dynamometer from April 2016 to June 2017. | 15 months
  Evaluate the incidence of OTAGO's physical intervention program on improvement of parameters of physical frailty (endurance) in elderly (75-89years). Starting training with phase guided by physiotherapist, followed by loyalty phase guided by regular nurse. It will be tested as strength measured with dynamometer in leg and arm. It will be monitoring at baseline and during follow-up.
Appointment at the surgery measured through questionnaire of number of appointment in the practice | 15 months
  Evaluate the incidence of OTAGO's physical intervention program on reduction of appointment in the practice of primary and second care and hospital admission in elderly (75-89years). Starting training with phase guided by physiotherapist, followed by loyalty phase guided by regular nurse. It will be measured through questionnaire of number of appointment in the practice in the previous year and during follow-up.
Nursing Home admittance measured through questionnaire | 15 months
  Evaluate the incidence of OTAGO's physical intervention program on reduction of inclusion rate in home care or institutionalization in elderly (75-89years). Starting training with phase guided by physiotherapist, followed by loyalty phase guided by regular nurse. It will be measured through questionnaire of home care and/or institutionalization in the previous year and during follow-up.
Drug reduction measured through questionnaire of kind of drug from April 2016 to June 2017. | 15 months
  Evaluate the effect of drug reduction in the intervention of disprescription performed in the cohort by the usual care team in elderly (75-89 years). It will be measured through questionnaire of kind of drug, if there are any removed drug, and number and kind of drug removed to the end. Monitoring at baseline and during follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Azagra, PhD, Principal Investigator — Insitut Català de la Salut, Universitat Autònoma de Barcelona
Locations (11):
- Spain (11):
  - CAP Barberà del Vallès, Barbera Del Valles, Barcelona
  - CAP Canaletes, Cerdanyola del Vallès, Barcelona
  - CAP Serraparera, Cerdanyola del Vallès, Barcelona
  - CAP Creu Alta, Sabadell, Barcelona
  - CAP Badia del Vallés, Barcelona
  - CAP Castellar, Castellar del Vallès
  - CAP La Llagosta, La Llagosta
  - Cap Centre, Sabadell
  - Cap Can Rull, Sabadell
  - CAP Ca N'Oriach, Sabadell
  - CAP Sud, Sabadell

IPD SHARING:
Plan to Share IPD: Undecided